CLINICAL TRIAL: NCT07185698
Title: UVASC Urethral Vascularization and Urodynamics
Brief Title: Urethral Vascularization and Urodynamics
Acronym: UVASC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Diana Höhn, MD, Insel Gruppe AG, University Hospital Bern
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-01776; 2024-01776 (Other: Ethikkommission Bern)
Record Dates: First submitted 2025-09-04; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Stress Urinary Incontinence; Ultrasound; Vascularisation; Urodynamic Exam
MeSH Terms: conditions — Urinary Incontinence, Stress; Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress urinary incontinence (Experimental): participants with stress urinary incontinence
  Interventions: Diagnostic Test: 3D Ultrasound
- NO Stress Urinary Incontinence (Experimental): Participants referred to urodynamics without stress urinary incontinence
  Interventions: Diagnostic Test: 3D Ultrasound

INTERVENTIONS:
Diagnostic Test: 3D Ultrasound — Virtual Organ Computer-aided AnaLysis (VOCAL) to assess flow and velocity characteristics of the urethral blood supply

SUMMARY:
The urethra plays a crucial role in maintaining urinary continence. Its complex blood supply is still not well understood. Particularly in the context of urethral pressure. Urethral pressure can be measured by bladder and urethral pressure studies (urodynamic).

This study aims to use advanced imaging techniques to analyse the blood supply of the urethra and correlate it to urethral pressure measurements.

Elucidating these relationships will improve our understanding of urethral function and malfunction, and ultimately optimise diagnosis and treatment of stress urinary incontinence. A total of 35 participants with stress urinary incontinence and 35 without stress urinary incontinence will be asked to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Urodynamic examination
* Written informed consent
* Understanding of the German language
* Indicated urodynamic assessment
* Endovaginal and perineal ultrasound feasible

Exclusion Criteria:

* Urinary tract infections
* Transgender Population
* Pregnancy
* History of incontinence or prolapse surgery
* Pelvic prolapse higher than second degree
* Prior pelvic radiotherapy
* Prior history of gynecologic tumor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Color histogram index (Vascularity Index) | Enrollment by the urodynamic examination until the ultrasound measurement (VOCAL) up to 4 weeks
  Doppler Indices (Vascularity Index) generated by Virtual Organ Computer-aided AnaLysis (VOCAL)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Hoehn, MD, Principal Investigator — Women's Hospital, University Hospital Bern, Inselspital, Switzerland
Locations (1):
- University Hospital Bern, Inselspital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
According to the ethics application, the confidentiality measures of the study do not allow the public release of participant data. However, data can be made available upon reasonable request.

REFERENCES:
- [Background] Lone F, Thakar R, Wieczorek AP, Sultan AH, Stankiewicz A. Assessment of urethral vascularity using 2D colour Doppler high-frequency endovaginal ultrasonography in women treated for symptomatic stress urinary incontinence: 1-year prospective follow-up study. Int Urogynecol J. 2016 Jan;27(1):85-92. doi: 10.1007/s00192-015-2800-z. Epub 2015 Aug 5. PMID 26243181
- [Background] Liang CC, Chang SD, Chang YL, Wei TY, Wu HM, Chao AS. Three-dimensional power Doppler measurement of perfusion of the periurethral tissue in incontinent women -- a preliminary report. Acta Obstet Gynecol Scand. 2006;85(5):608-13. doi: 10.1080/00016340500342920. PMID 16752242
- See also: UniBE Forschungsstiftung Grant — https://forschungsstiftung.ch/wp-content/uploads/2025/06/Jahresbericht-2024-UBFS.pdf
- See also: Grant from the Burgergemeinde Bern — https://www.bgbern.ch/themen/engagements/wissenschaftsfoerderung
- See also: Grant from Vontobel Stiftung — https://www.vontobel-stiftung.ch/de-ch/
- See also: Grant from Ruth und Arthur Scherbarth Stiftung — https://boris-portal.unibe.ch/entities/funding/2f916336-712d-47da-aaba-39e2a61eafc8